CLINICAL TRIAL: NCT02702388
Title: A Multicenter, Randomized, Double-Blind Phase 2 Trial of Lenvatinib (E7080) in Subjects With 131I-Refractory Differentiated Thyroid Cancer to Evaluate Whether an Oral Starting Dose of 18 mg Daily Will Provide Comparable Efficacy to a 24-mg Starting Dose, But Have a Better Safety Profile
Brief Title: A Trial of Lenvatinib (E7080) in Subjects With Iodine-131 Refractory Differentiated Thyroid Cancer to Evaluate Whether an Oral Starting Dose of 18 Milligram (mg) Daily Will Provide Comparable Efficacy to a 24 mg Starting Dose, But Have a Better Safety Profile
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E7080-G000-211; 2014-005199-27 (EudraCT Number)
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2020-12

CONDITIONS: Thyroid Cancer
Keywords: Lenvatinib; E7080; Iodine-131 Refractory Differentiated Thyroid Cancer; Lenvima; Phase 2; RR-DTC
MeSH Terms: conditions — Thyroid Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 24 mg Lenvatinib (Experimental): Participants will receive 24 mg once daily (QD) as the starting dose. Dose reductions will occur in succession based on the previous dose level (24, 20, 14, 10, or 8 mg QD). To maintain blinded treatment assignment, participants will be administered study drug in the form of two 10-mg capsules and two 4-mg capsules containing either lenvatinib or placebo (total of 4 capsules) to be taken orally, at approximately the same time each morning and may be taken in a fasting state or following a meal.
  Interventions: Drug: Lenvatinib; Drug: Lenvatinib matching placebo
- 18 mg Lenvatinib (Experimental): Participants will receive 18mg QD as the starting dose. Dose reductions will occur in succession based on the previous dose level (18,14, 10, 8, or 4 mg QD). To maintain blinded treatment assignment, participants will be administered study drug in the form of two 10-mg capsules and two 4-mg capsules containing either lenvatinib or placebo (total of 4 capsules) to be taken orally, at approximately the same time each morning and may be taken in a fasting state or following a meal.
  Interventions: Drug: Lenvatinib; Drug: Lenvatinib matching placebo

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsule.
  Other Names: Lenvima; E7080
Drug: Lenvatinib matching placebo — Lenvatinib matching placebo capsule.

SUMMARY:
This is a multicenter, randomized, double-blind study being conducted as a postmarketing requirement to the US Food and Drug Administration (FDA) to evaluate whether there is a lower starting dosage of lenvatinib 24 mg once daily (QD) that provides comparable efficacy but has a better safety profile in participants with radioiodine-refractory differentiated thyroid cancer RR-DTC with radiographic evidence of disease progression within the prior 12 months.

DETAILED DESCRIPTION:
This study consists of 2 phases, the Prerandomization Phase and the Randomization Phase. The Prerandomization Phase will last no longer than 28 days and will include a Screening Period to establish protocol eligibility and a Baseline Period to confirm eligibility and establish disease characteristics prior to randomization and treatment.

The Randomization Phase will consist of a Treatment Period and a Follow-up Period. It will begin at the time of randomization of the first participant and will consist of 28-day blinded study treatment cycles. The data cutoff for the primary analysis will occur at the end of the Randomization Phase, which is defined as when the last participant enrolled completes the Week 24 tumor assessments or discontinues study treatment if before Week 24.

Participants on treatment at the time of data cutoff for the primary analysis will remain on blinded investigational product until the primary analysis has been completed, after which they will transition to commercial lenvatinib outside the study. The last participant's last assessment (Off-treatment visit) will be the End of Study.

Participants will be randomly assigned to treatment with 1 of 2 blinded starting dosages of lenvatinib in a 1:1 ratio to receive lenvatinib 18 mg or 24 mg orally once daily (QD). Dose reductions will occur in succession based on the previous dose level (24, 20, 14, 10, and 8 mg QD, or 18, 14, 10, 8, and 4 mg QD, respectively). Once the dose has been reduced, it may not be increased at a later date.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed diagnosis of one of the following differentiated thyroid cancer (DTC) subtypes:

   1. Papillary thyroid cancer (PTC)

      * Follicular variant
      * Variants (including but not limited to tall cell, columnar cell, cribriform-morular, solid, oxyphil, Warthin's-like, trabecular, tumor with nodular fasciitis-like stroma, Hürthle cell variant of papillary carcinoma, poorly differentiated)
   2. Follicular thyroid cancer (FTC)

      * Hurthle cell
      * Clear cell
      * Insular
2. Measurable disease meeting the following criteria and confirmed by central radiographic review:

   1. At least 1 lesion of greater than or equal to (>=)1.0 centimeter (cm) in the longest diameter for a non-lymph node or >=1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) using computed tomography/magnetic resonance imaging (CT/MRI). If there is only 1 target lesion and it is a non-lymph node, it should have a longest diameter of >=1.5 cm.
   2. Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
3. Participants must show evidence of disease progression within 12 months (an additional month will be allowed to accommodate actual dates of performance of screening scans, that is, within less than or equal to <=13 months) prior to signing informed consent, according to RECIST 1.1 assessed and confirmed by central radiographic review of CT and/or MRI scans.
4. Participants must be Iodine-131 refractory/resistant as defined by at least one of the following:

   1. One or more measurable lesions that do not demonstrate iodine uptake on any radioiodine scan.
   2. One or more measurable lesions that have progressed according to RECIST 1.1 within 12 months (an additional month will be allowed to accommodate actual dates of performance of screening scans, ie, within ≤13 months) after Iodine-131 therapy, despite demonstration of radioiodine avidity at the time of that treatment by pre- or posttreatment scanning. These participants must not be eligible for possible curative surgery.
   3. Cumulative activity of Iodine-131 of greater than (>) 600 millicurie (mCi) or 22 gigabecquerels (GBq), with the last dose administered at least 6 months prior to study entry.
5. Participants with known brain metastases who have completed whole brain radiotherapy, stereotactic radiosurgery or complete surgical resection, will be eligible if they have remained clinically stable, asymptomatic, and off steroids for one month.
6. Participants must be receiving thyroxine suppression therapy and thyroid stimulating hormone (TSH) should not be elevated (TSH should be <=5.50 micro-international units per liter [mcIU/ML]). When tolerated by the participant, thyroxine dose should be changed to achieve TSH suppression (TSH <0.50 mcIU/ML) and this dose may be changed concurrently upon starting study drug treatment.
7. All chemotherapy or radiation-related toxicities must have resolved to Grade <2 severity per Common Terminology Criteria for Adverse Events (CTCAE v4.03), except alopecia and infertility.
8. Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
9. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mmHg at Screening and no change in antihypertensive medications within 1 week prior to Cycle 1/Day 1.
10. Adequate renal function defined as calculated creatinine clearance >=30 mL/min per the Cockcroft and Gault formula.
11. Adequate bone marrow function:

    1. Absolute neutrophil count (ANC) >=1500/mm^3 (>=1.5*10^3/uL)
    2. Platelets >=100,000/mm^3 (>=100*10^9/L)
    3. Hemoglobin >=9.0 g/dL
12. Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) <=1.5.
13. Adequate liver function:

    1. Bilirubin <=1.5*upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome.
    2. Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <=3*ULN (<=5*ULN if participant has liver metastases). If alkaline phosphatase is >3*ULN (in absence of liver metastases) or >5*ULN (in presence of liver metastases) AND the participant also is known to have bone metastases, the liver-specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of total alkaline phosphatase.
14. Males or females age >=18 years at the time of informed consent.
15. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of B-hCG. A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
16. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least 1 month before dosing).
17. Females of childbearing potential should avoid becoming pregnant and use highly effective contraception while on treatment with lenvatinib and for at least 1 month after finishing treatment. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (example, total abstinence, an intrauterine device, a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation. Women using oral hormonal contraceptives should add a barrier method.
18. Participants must voluntarily agree to provide written informed consent.
19. Participants must be willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Anaplastic or medullary carcinoma of the thyroid.
2. Diagnosed with meningeal carcinomatosis.
3. Two or more prior vascular endothelial growth factor (VEGF)/vascular endothelial growth factor receptor (VEGFR)-targeted therapies or any ongoing treatment for RR-DTC other than TSH-suppressive thyroid hormone therapy.
4. Prior treatment with lenvatinib.
5. Participants who have received any anticancer treatment within 21 days or any investigational agent within 30 days (or 5 half-lives) prior to the first dose of study drug and should have recovered from any toxicity related to previous anticancer treatment. This does not apply to the use of TSH suppressive thyroid hormone therapy.
6. Major surgery (example, laparotomy, thoracotomy or joint replacement) within 3 weeks prior to randomization or elective surgery scheduled to be performed during the study.
7. Participants having >1+ proteinuria on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein >=1 g/24 h will be ineligible.
8. Gastrointestinal malabsorption or any other condition that in the opinion of the investigator might affect the absorption of study drug.
9. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or cerebral vascular accident within 6 months of the first dose of study drug, or cardiac arrhythmia associated with hemodynamic instability.
10. Prolongation of corrected QT interval (QTc) to >480 ms as demonstrated by a repeated electrocardiogram (ECG) or a clinically significant ECG abnormality, including a marked prolonged QT/QTc interval (example, a repeated demonstration of a QTc interval >500 ms).
11. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
12. Active infection (any infection requiring treatment).
13. Active malignancy (except for DTC or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months.
14. Bleeding or thrombotic disorders.
15. Known intolerance to study drug (or any of the excipients).
16. Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study.
17. Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (101):
- United States (16):
  - Facility#1, La Jolla, California
  - Facility #1, San Diego, California
  - Facility #1, Torrance, California
  - Facility #1, Washington D.C., District of Columbia
  - Facility #1, Boston, Massachusetts
  - Facility #2, Boston, Massachusetts
  - Facility #1, Ann Arbor, Michigan
  - Facility #1, Detroit, Michigan
  - Facility#2, Morristown, New Jersey
  - Facility#1, Summit, New Jersey
  - Facility #1, The Bronx, New York
  - Facility #1, Columbus, Ohio
  - Facility #1, Portland, Oregon
  - Facility #2, Philadelphia, Pennsylvania
  - Facility #1, Philadelphia, Pennsylvania
  - Facility #1, Seattle, Washington
- Australia (9):
  - Facility #1, Darlinghurst, New South Wales
  - Facility #1, Saint Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Facility#2, Chermside, Queensland
  - Facility #1, Herston, Queensland
  - Facility #1, Melbourne, Victoria
  - Facility #1, Nedlands, Western Australia
  - Facility #1, Melbourne
  - Facility #1, Saint Leonards
- Belgium (4):
  - Facility #1, Edegem, Antwerpen
  - Facility #1, Brussels, Brussels Capital
  - Facility #2, Namur
  - Facility #1, Namur
- Canada (3):
  - Facility #1, Calgary, Alberta
  - Facility #1, Toronto, Ontario
  - Facility #1, Québec
- Facility #1, Odense, Region Syddanmark, Denmark
- France (13):
  - Facility #1, Strasbourg, Bas-Rhin
  - Facility #1, Caen, Calvados
  - Facility #1, Dijon, Cote-d'Or
  - Facility #1, Bordeaux, Gironde
  - Facility #1, Angers, Maine-et-Loire
  - Facility #2, Villejuif, Val-de-Marne
  - Facility #1, Villejuif, Val-de-Marne
  - Facility #2, Angers
  - Facility #1, Bordeaux
  - Facility #1, Caen
  - Facility #1, Dijon
  - Facility #2, Lyon
  - Facility #1, Paris
- Germany (7):
  - Facility #1, Tübingen, Baden-Wurttemberg
  - Facility #1, Würzburg, Bavaria
  - Facility #1, Hanover, Lower Saxony
  - Facility #1, Essen, North Rhine-Westphalia
  - Facility #2, Essen, North Rhine-Westphalia
  - Facility #1, Essen
  - Facility #1, Leipzig
- Facility #1, Petah Tikva, Israel
- Italy (17):
  - Facility #6, Rome, Lazio
  - Facility #1, Rome, Lazio
  - Facility #2, Rome, Lazio
  - Facility #3, Rome, Lazio
  - Facility #2, Milan, Lombardy
  - Facility #3, Milan, Lombardy
  - Facility #4, Milan, Lombardy
  - Facility #5, Milan, Lombardy
  - Facility #1, Livorno, Tuscany
  - Facility #1, Pisa, Tuscany
  - Facility #6, Milan
  - Facility #7, Milan
  - Facility #2, Pisa
  - Facility #4, Roma
  - Facility #2, Rozzano
  - Facility #1, Torino
  - Facility #1, Viagrande
- Facility #2, Kielce, Poland
- Romania (2):
  - Facility #1, Cluj-Napoca, Cluj
  - Facility #1, Bucharest
- Russia (9):
  - Facility #4, Saint Petersburg, Leningradskaya O
  - Facility #3, Moscow
  - Facility #4, Moscow
  - Facility #1, Moscow
  - Facility #2, Moscow
  - Facility #1, Obninsk
  - Facility #3, Saint Petersburg
  - Facility #1, Saint Petersburg
  - Facility #2, Saint Petersburg
- South Korea (6):
  - Facility#1, Busan
  - Facility #1, Goyang-si
  - Facility #3, Seoul
  - Facility #4, Seoul
  - Facility #1, Seoul
  - Facility #2, Seoul
- Spain (8):
  - Facility #1, Barcelona, Catalonia
  - Facility #2, Madrid, Madrid, Communidad Delaware
  - Facility #1, Badalona
  - Facility #2, Barcelona
  - Facility #1, Madrid
  - Facility #2, Madrid
  - Facility #3, Madrid
  - Facility #1, Málaga
- Sweden (2):
  - Facility #1, Gothenburg
  - Facility #1, Lund
- United Kingdom (2):
  - Facility #1, London, City of London
  - Facility #1, Glasgow, Glasgow City

REFERENCES:
- [Derived] Taylor MH, Leboulleux S, Panaseykin Y, Konda B, de La Fouchardiere C, Hughes BGM, Gianoukakis AG, Park YJ, Romanov I, Krzyzanowska MK, Garbinsky D, Sherif B, Pan JJ, Binder TA, Sauter N, Xie R, Brose MS. Health-related quality-of-life analyses from a multicenter, randomized, double-blind phase 2 study of patients with differentiated thyroid cancer treated with lenvatinib 18 or 24 mg/day. Cancer Med. 2023 Feb;12(4):4332-4342. doi: 10.1002/cam4.5308. Epub 2022 Dec 4. PMID 36464853
- [Derived] Brose MS, Panaseykin Y, Konda B, de la Fouchardiere C, Hughes BGM, Gianoukakis AG, Joo Park Y, Romanov I, Krzyzanowska MK, Leboulleux S, Binder TA, Dutcus C, Xie R, Taylor MH. A Randomized Study of Lenvatinib 18 mg vs 24 mg in Patients With Radioiodine-Refractory Differentiated Thyroid Cancer. J Clin Endocrinol Metab. 2022 Feb 17;107(3):776-787. doi: 10.1210/clinem/dgab731. PMID 34664662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 38 investigative sites in the North America, Europe, Russia, Australia, and Asia. As planned, the study was unblinded after the primary analysis was completed and all participants were treated with open-label lenvatinib at their current dose level at the discretion of the investigator until they were transitioned to commercially available lenvatinib.
Pre-assignment Details: A total of 241 participants were screened and enrolled of which 89 participants were screen failures, and 152 participants were randomized and treated.
Groups:
- Lenvatinib 24 mg: Participants received lenvatinib 24 mg, capsule, orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first (up to 35 months). To maintain blinded treatment assignment, participants received a total of 4 capsules in the form of two 10-mg capsules and one 4-mg capsule containing lenvatinib and one 4-mg placebo capsule.
- Lenvatinib 18 mg: Participants received lenvatinib 18 mg, capsule, orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first (up to 35 months). To maintain blinded treatment assignment, participants received a total of 4 capsules in the form of one 10-mg capsule and two 4-mg capsules containing lenvatinib and one 10-mg placebo capsule.
Period: Overall Study
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Started | 75 | 77
Completed | 35 | 26
Not Completed | 40 | 51
Not completed — Disease Progression | 18 | 25
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Adverse Event | 11 | 15
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants randomly assigned to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg | Total
Number analyzed (Participants) | 75 | 77 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.58) | 64.4 (11.79) | 64.4 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 40 | 74
  Male | 41 | 37 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 71 | 67 | 138
  Unknown or Not Reported | 1 | 6 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 11 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 46 | 40 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 23 | 38

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as of Week 24 (ORR24wk)
Description: ORR as of Week 24 was defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) as of the Week 24 time point or earlier, as measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). PR: was at least a 30 percent (%) decrease in sum of diameter (SOD) of target lesions, taking as reference the baseline SOD.
Time Frame: From the date of randomization up to Week 24
Population: FAS included all participants randomly assigned to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
percentage of participants | 57.3 [46.1 to 68.5] | 40.3 [29.3 to 51.2]
Statistical Analysis 1: Comparison: Lenvatinib 24 mg vs Lenvatinib 18 mg; Test type: Non-Inferiority — Odds ratio of ORR as of Week 24 response (18 mg vs 24 mg) along with its 95% confidence interval (CI) using the Cochran-Mantel-Haenszel (CMH) method, stratified by the randomization stratification factors. The test was performed per the 95% CI using the noninferiority margin of 0.4. Noninferiority will be declared if the lower limit of the 95% CI for the odds ratio is greater than 0.4; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.26 to 0.96]

2. Primary Outcome: Percentage of Participants With Grade 3 or Higher Treatment-emergent Adverse Events (TEAEs) in the First 24 Weeks
Description: This outcome measure reports TEAEs in the first 24 weeks only. A TEAE was defined as any adverse event (AE) that had an onset date on or after the first dose of study drug up to 28 days following the last dose of study drug, or a worsening in severity from Baseline (pretreatment). In addition, if an AE reemerged during treatment, having been present at pretreatment (Baseline) but stopped before treatment, it was also counted as a TEAE. A severity grade was defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. As per CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Time Frame: Baseline up to Week 24
Population: Safety analysis set included all participants randomly assigned to treatment and who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
percentage of participants | 61.3 | 57.1

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS, defined as the time from the date of randomization to the date of first documentation of PD, or date of death, whichever occurs first, as measured by RECIST V1.1. PD: 20% increase in the sum of the pertinent diameters (SOD) of target lesions, taking as reference the smallest sum SOD recorded since the treatment started or the appearance of one or more new lesions. PFS was analyzed using the Kaplan-Meier method. As planned, data for this endpoint was analyzed and collected till Primary completion date.
Time Frame: Time from the date of randomization to the date of first documentation of PD, or date of death, whichever occurs first up to approximately 2 years 6 months
Population: FAS included all participants randomly assigned to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
months | NA [22.1 to NA] — Median and maximum range of 95% CI was not estimable because insufficient number of participants had events. | 24.4 [14.7 to NA] — Maximum range of 95% CI was not estimable because insufficient number of participants had events.

4. Secondary Outcome: PFS After Next Line of Treatment (PFS2)
Description: PFS2, defined as the time from randomization to PD on next-line treatment, or death from any cause, whichever occurred first, as measured by RECIST V1.1. PD: 20% increase in the SOD of target lesions, taking as reference the smallest sum SOD recorded since the treatment started or the appearance of one or more new lesions. PFS was analyzed using the Kaplan-Meier method. As planned, data for this endpoint was analyzed and collected till Primary completion date.
Time Frame: Time from randomization to PD on next-line treatment or death from any cause, whichever occurs first up to approximately 2 years 6 months
Population: FAS included all participants randomly assigned to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
months | NA [NA to NA] — Median and 95% CI was not estimable because insufficient number of participants had events. | NA [22.1 to NA] — Median and maximum range of 95% CI was not estimable because insufficient number of participants had events.

5. Secondary Outcome: Number of Participants With TEAE and Serious Adverse Events (SAEs)
Description: TEAEs were defined as those AEs that occurred (or worsened, if present at Baseline) after the first dose of study drug through 28 days after the last dose of study drug. An AE was defined as any untoward medical occurrence in a participants or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. SAE was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect.
Time Frame: From date of first administration of study drug up to 28 days after last dose of study drug up to approximately 3 years 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
Participants
  TEAE | 75 | 76
  SAE | 26 | 35

6. Secondary Outcome: Time to Treatment Discontinuation Due to an Adverse Event (AE)
Description: Time to Treatment Discontinuation due to an AE (such as abdominal distention, appendicitis perforated, arthralgia, anemia, etc) was analyzed using the Kaplan-Meier method. As planned, data for this endpoint was analyzed and collected till Primary completion date.
Time Frame: From date of first administration of study drug up to approximately 2 years 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
weeks | NA [NA to NA] — Median and 95% CI were not estimable because insufficient number of participants had events. | NA [84.3 to NA] — Median and maximum range of 95% CI were not estimable because insufficient number of participants had events.

7. Secondary Outcome: Number of Dose Reductions
Description: Number of dose reduction was reported as number of participants who underwent one or more number of dose reductions. As planned, data for this endpoint was analyzed and collected till Primary completion date.
Time Frame: From date of first administration of study drug up to approximately 2 years 6 months
Population: Safety analysis set included all participants randomly assigned to treatment and who received at least 1 dose of study drug. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 53 | 45
Participants
  1 Dose Reduction | 17 | 20
  2 Dose Reduction | 20 | 13
  3 Dose Reduction | 13 | 8
  greater than or equal to (>=) 4 Dose Reduction | 3 | 4

8. Secondary Outcome: Time to First Dose Reduction
Description: Time to First Dose Reduction was analyzed using the Kaplan-Meier method. As planned, data for this endpoint was analyzed and collected till Primary completion date.
Time Frame: From date of first administration of study drug up to approximately 2 years 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
weeks | 15.3 [12.1 to 20.1] | 24.1 [11.1 to 35.9]

9. Secondary Outcome: Model Predicted Apparent Total Clearance (CL/F) Following Oral Dosing of Lenvatinib
Description: Sparse pharmacokinetic (PK) samples (approximately 9 per participant) were collected and analyzed using a population PK approach to estimate PK parameters. Lenvatinib total plasma concentration data were pooled with data from studies E7080-G000-303 (NCT01321554) and E7080-G000-201 (NCT00784303), and a population PK model was applied to the pooled dataset. Individual predicted CL/F for lenvatinib was then derived from the PK model by starting dose.
Time Frame: Cycle 1 Day 1: 0.5-4 hours and 6-10 hours postdose; Cycle 1 Day 8: predose, Cycle 1 Day 15: predose, 0.5-4 hours and 6-10 hours postdose; Cycle 1 Day 22: optionally at predose; Cycle 2 Day 1: predose and 2-12 hours postdose (Cycle length=28 days)
Population: PK Analysis Set included all participants who received at least one dose of study drug and who had evaluable lenvatinib plasma concentration data. Population for Lenvatinib 24 mg arm for this outcome measure included participants from study E7080-G000-303 (NCT01321554), E7080-G000-201 (NCT00784303) and from this current study E7080-G000-211. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Groups:
- Lenvatinib 24 mg: All participants received lenvatinib 24 mg, capsule orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first in studies E7080-G000-303 (NCT01321554), E7080-G000-201 (NCT00784303) and this current study (E7080-G000-211).
- Lenvatinib 18 mg: Participants received lenvatinib 18 mg, capsule, orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first (up to 35 months) in this current study E7080-G000-211. To maintain blinded treatment assignment, participants received a total of 4 capsules in the form of one 10-mg capsule and two 4-mg capsules containing lenvatinib and one 10-mg placebo capsule.
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 439 | 73
liter per hour (L/h) | 6.408 (1.945) | 6.243 (2.278)

10. Secondary Outcome: Model Predicted Area Under the Plasma Drug Concentration-time Curve (AUC) for Lenvatinib
Description: Sparse PK samples (approximately 9 per participant) were collected and analyzed using a population PK approach to estimate PK parameters. Lenvatinib total plasma concentration data were pooled with data from studies E7080-G000-303 (NCT01321554) and E7080-G000-201 (NCT00784303), and a population PK model was applied to the pooled dataset. Individual predicted AUC for lenvatinib was then derived from the PK model by starting dose.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 439 | 73
nanogram*hour per milliliter (ng*h/mL) | 3747 (1295) | 3370 (4438)

11. Secondary Outcome: Parameter Estimates From the Population Pharmacokinetic/Pharmacodynamic (PK/PD) Model Describing the Relationship Between Lenvatinib Exposure (AUC) and Thyroglobulin Levels
Description: The relationship between exposure to lenvatinib and change from baseline in thyroglobulin was planned to be analyzed using a model-based approach.
Time Frame: as for outcome 9
Population: PK/PD modeling of the effect of lenvatinib exposure on thyroglobulin levels could not be achieved due to the high variability in change from baseline data and hence data was not collected and reported.
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Parameter Estimates From the Population Pharmacokinetic/Pharmacodynamic (PK/PD) Model Describing the Relationship Between Lenvatinib Exposure (AUC) and Thyroid-Stimulating Hormone (TSH) Levels
Description: The relationship between exposure to lenvatinib and change from baseline in TSH was planned to be analyzed using a model-based approach.
Time Frame: as for outcome 9
Population: PK/PD modeling of the effect of lenvatinib exposure on TSH levels could not be achieved due to the high variability in change from baseline data and hence data was not collected and reported.
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Baseline Level Estimates From the Population PK/PD Model Describing the Relationship Between Lenvatinib Exposure (AUC) and Vascular Endothelial Growth Factor (VEGF), Soluble Tie-2, Angiopoietin-2 (Ang-2) and Fibroblast Growth Factor-23 (FGF23) Levels
Description: Per the planned population PK/PD analysis for this endpoint, Arms/Groups were combined and lenvatinib total plasma concentration and serum biomarker data for VEGF, Ang-2, soluble Tie-2, and FGF23 from this study were combined with data from study E7080-G000-303 (NCT01321554). The relationship between lenvatinib exposure at the time of measurement of biomarker was described using PK/PD modelling. Initially, PK/PD models were developed individually for each biomarker and then combined into a single combined model. Changes in biomarker levels over time related to lenvatinib exposure were best described by an indirect response, sigmoidal Emax model. For the final combined model, baseline level estimates were determined separately for each biomarker. The data presented are the model predicted baseline estimates, with Measure Type "Number." They are population PK/PD model predictions and have been estimated using non-linear mixed effects modelling.
Time Frame: as for outcome 9
Population: PK/PD analysis was performed for differentiated thyroid cancer (DTC) participants who received lenvatinib or placebo in study E7080-G000-303 (NCT01321554) and current study E7080-G000-211 and provided both PK data for lenvatinib and baseline and post-dose serum biomarkers samples. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for given categories.
Measure: Number (95% Confidence Interval); unit: nanogram per liter (ng/L)
Groups:
- Lenvatinib or Placebo - All Participants: All participants who received lenvatinib 24 mg or 18 mg or placebo, capsule, orally, once daily in a 28-day treatment cycles until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first in studies E7080-G000-303 (NCT01321554) and this current study (E7080-G000-211).
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 560
nanogram per liter (ng/L)
  VEGF | 0.370 [0.355 to 0.385]
  Tie-2 | 14.6 [14.4 to 14.8]
  Ang-2 | 3.36 [3.26 to 3.46]
  FGF23: number analyzed (Participants) | 542
  FGF23 | 0.0990 [0.0949 to 0.103]

14. Secondary Outcome: Mean Residence Time (MRT) Estimates From the Population PK/PD Model Describing the Relationship Between Lenvatinib Exposure (AUC) and VEGF, Soluble Tie-2, Ang-2 and FGF23 Levels
Description: Per the planned population PK/PD analysis for this endpoint, Arms/Groups were combined and lenvatinib total plasma concentration and serum biomarker data for VEGF, Ang-2, soluble Tie-2, and FGF23 from this study were combined with data from study E7080-G000-303 (NCT01321554). The relationship between lenvatinib exposure at the time of measurement of biomarker was described using PK/PD modelling. Initially, PK/PD models were developed individually for each biomarker and then combined into a single combined model. Changes in biomarker levels over time related to lenvatinib exposure were best described by an indirect response, sigmoidal Emax model. For the final combined model, MRT estimates were determined separately for each biomarker. The data presented are the model predicted MRT estimates, with Measure Type "Number." They are population PK/PD model predictions and have been estimated using non-linear mixed effects modelling.
Time Frame: as for outcome 9
Population: PK/PD analysis was performed for DTC participants who received lenvatinib or placebo in study E7080-G000-303 (NCT01321554) and current study E7080-G000-211 and provided both PK data for lenvatinib and baseline and post-dose serum biomarkers samples. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for given categories.
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 560
hours
  VEGF | 58.3 [23.4 to 93.2]
  Tie-2 | 354 [314 to 394]
  Ang-2 | 173 [134 to 212]
  FGF23: number analyzed (Participants) | 542
  FGF23 | 265 [185 to 345]

15. Secondary Outcome: Hill Coefficient Estimates From the Population PK/PD Model Describing the Relationship Between Lenvatinib Exposure (AUC) and VEGF, Soluble Tie-2, Ang-2 and FGF23 Levels
Description: Per the planned population PK/PD analysis for this endpoint, Arms/Groups were combined and lenvatinib total plasma concentration and serum biomarker data for VEGF, Ang-2, soluble Tie-2, and FGF23 from this study were combined with data from study E7080-G000-303 (NCT01321554). The relationship between lenvatinib exposure at the time of measurement of biomarker was described using PK/PD modelling. Initially, PK/PD models were developed individually for each biomarker and then combined into a single combined model. Changes in biomarker levels over time related to lenvatinib exposure were best described by an indirect response, sigmoidal Emax model. For the final combined model, Hill Coefficient estimates were determined separately for each biomarker. The data presented are the model predicted Hill Coefficient estimates, with Measure Type "Number." They are population PK/PD model predictions and (&) have been estimated using non-linear mixed effects modelling.
Time Frame: as for outcome 9
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: unitless
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 560
unitless
  VEGF | 1.00 [NA to NA] — Upper and lower 95% CI was not estimable since Hill coefficient was fixed to 1 as the model was unstable. Hence, the CI was not estimated and reported.
  Tie-2 | 0.313 [0.242 to 0.384]
  Ang-2 | 4.27 [2.92 to 5.62]
  FGF23: number analyzed (Participants) | 542
  FGF23 | 1.00 [NA to NA] — Upper and lower 95% CI was not estimable since Hill coefficient was fixed to 1 as the model was unstable. Hence, the CI was not estimated and reported.

16. Secondary Outcome: Parameter Estimates From the PK/PD Model for Tumor Growth Inhibition and Serum Biomarkers Tie-2 and Ang-2
Description: Per the planned analysis, Arms/Groups were combined & tumor-growth inhibition models based on lenvatinib & placebo data from this study combined with study NCT01321554. Effects of tumor growth rate, drug effects, tumor resistance, & tumor size reduction related to biomarker response were assessed. Longitudinal data of sum of the longest diameter for target lesion by investigator assessment in this study & independent reviewer assessment in study NCT01321554 were used. Changes in Ang-2 & soluble Tie-2 were evaluated, individually & in combination for their impact on tumor size. The concomitant use of lenvatinib & biomarker changes due to drug effects as predictors of tumor size were also evaluated. The final integrated model for tumor growth & biomarkers included effects of lenvatinib exposure & tumor growth reduction related to Tie-2 & Ang-2 biomarkers as significant predictors. Data presented are the parameters defining this non-linear mixed effects model, with Measure Type "Number."
Time Frame: Baseline up to week 120
Population: PK/PD analysis was performed for DTC participants who received lenvatinib or placebo in study E7080-G000-303 (NCT01321554) and this current study E7080-G000-211 who had PK data and at least one post-baseline tumor evaluation. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: per week
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 558
per week
  Tumor growth rate | 0.00249 [0.00177 to 0.00321]
  Maximum effect of lenvatinib on tumor suppression (Emax) | 0.0877 [0.0843 to 0.0911]
  Resistance term | 0.268 [0.253 to 0.283]
  Tumor size reduction rate constant for Tie-2 | -0.0220 [-0.0247 to 0.0193]
  Tumor size reduction rate constant for Ang-2 | -0.0146 [-0.0158 to -0.0134]

17. Secondary Outcome: Lenvatinib Mean AUC Resulting in 50% of the Emax (EC50) Estimate From the PK/PD Model for Tumor Growth Inhibition and Serum Biomarkers Tie-2 and Ang-2
Description: Per the planned analysis, Arms/Groups were combined & tumor-growth inhibition models based on lenvatinib & placebo data from this study combined with study NCT01321554. Effects of tumor growth rate, drug effects, tumor resistance, & tumor size reduction related to biomarker response were assessed. Longitudinal data of the sum of the longest diameter for target lesion by investigator assessment in this study & independent reviewer assessment in study NCT01321554 were used. Changes in Ang-2 & soluble Tie-2 were evaluated, individually & in combination for their impact on tumor size. The concomitant use of lenvatinib & biomarker changes due to drug effects as predictors of tumor size were also evaluated. The final integrated model for tumor growth & biomarkers included effects of lenvatinib exposure & tumor growth reduction related to Tie-2 & Ang-2 biomarkers as significant predictors. Data presented are EC50 estimated using non-linear mixed effects modeling, with Measure Type "Number."
Time Frame: Baseline up to week 120
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: ng*h/mL
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 558
ng*h/mL | 1760 [1490 to 2030]

18. Secondary Outcome: Scale Factor Estimate for Final Parametric Time to Event PK/PD Model for PFS
Description: Per planned analysis, Arms/Groups were combined & PK/PD analysis for PFS was based on lenvatinib & placebo data from this study combined with NCT01321554. Relationship between lenvatinib exposure & PFS was assessed using Kaplan-Meier plots. A parametric survival model (proportional hazard model) with Weibull distribution structure was developed to estimate the probability distribution of time from study start to progression, as a function of covariates including baseline disease characteristics, demographics, lenvatinib exposure, changes in biomarker time profiles, model predicted change from baseline in tumor size & change in tumor size time-profiles. Significant (p<0.01) covariates from the univariate analysis were added to the model simultaneously & significant predictors were retained according to backward exclusion criteria (log likelihood ratio test, p-value of 0.001). Data presented are scale factor estimated using non-linear mixed effects modeling, with Measure Type "Number."
Time Frame: Time from the date of randomization to the date of first documentation of PD, or date of death, whichever occurred first up to approximately 3 years 3 months
Population: PK/PD analysis for PFS was performed for DTC participants who received lenvatinib or placebo in study E7080-G000-303 (NCT01321554) and this current study E7080-G000-211. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: per week
Groups:
- Lenvatinib or Placebo - All Participants: All participants received lenvatinib 24 mg or 18 mg or placebo, capsule orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first in studies E7080-G000-303 (NCT01321554) and this current study (E7080-G000-211).
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 475
per week
  Scale factor | 0.00700 [0.00353 to 0.0105]
  Scale factor drop out | 0.0000935 [0.000000188 to 0.000187]

19. Secondary Outcome: Shape Factor Estimate for Final Parametric Time to Event PK/PD Model for PFS
Description: Per planned analysis, Arms/Groups were combined & PK/PD analysis for PFS was based on lenvatinib & placebo data from this study combined with NCT01321554. Relationship between lenvatinib exposure & PFS was assessed using Kaplan-Meier plots. A parametric survival model (proportional hazard model) with Weibull distribution structure was developed to estimate the probability distribution of time from study start to progression, as a function of covariates including baseline disease characteristics, demographics, lenvatinib exposure, changes in biomarker time profiles, model predicted change from baseline in tumor size & change in tumor size time-profiles. Significant (p<0.01) covariates from the univariate analysis were added to the model simultaneously & significant predictors were retained according to backward exclusion criteria (log likelihood ratio test, p-value of 0.001). Data presented are shape factor estimated using non-linear mixed effects modeling, with Measure Type "Number."
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: unitless
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 475
unitless
  Shape factor | 1.36 [1.22 to 1.50]
  Shape factor drop out | 2.19 [1.96 to 2.42]

20. Secondary Outcome: Lenvatinib AUC Exposure Effect Estimate for Final Parametric Time to Event PK/PD Model for PFS
Description: Per planned analysis, Arms/Groups were combined & PK/PD analysis for PFS was based on lenvatinib & placebo data from this study combined with NCT01321554. Relationship between lenvatinib exposure & PFS was assessed using Kaplan-Meier plots. A parametric survival model (proportional hazard model) with Weibull distribution structure was developed to estimate probability distribution of time from study start to progression, as a function of covariates including baseline disease characteristics, demographics, lenvatinib exposure, changes in biomarker time profiles, model predicted change from baseline in tumor size & change in tumor size time-profiles. Significant (p<0.01) covariates from the univariate analysis were added to the model simultaneously & significant predictors retained according to backward exclusion criteria (log likelihood ratio test, p-value of 0.001). Data presented are AUC exposure effect estimated using non-linear mixed effects modeling, with Measure Type "Number."
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: per microgram*week per milliliter
Groups:
- Lenvatinib or Placebo - All Participants: All participants initially received lenvatinib 24 mg or 18 mg or placebo, capsule orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first in studies E7080-G000-303 (NCT01321554) and this current study (E7080-G000-211).
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 475
per microgram*week per milliliter | 0.00111 [0.000542 to 0.00168]

21. Secondary Outcome: Predicted Percent Change in Tumor Size Estimate for Final Parametric Time to Event PK/PD Model for PFS
Description: Per planned analysis, Arms/Groups were combined & PK/PD analysis for PFS based on lenvatinib & placebo data from this study combined with NCT01321554. Relationship between lenvatinib exposure & PFS was assessed using Kaplan-Meier plots. A parametric survival model (proportional hazard model) with Weibull distribution structure was developed to estimate probability distribution of time from study start to progression, as a function of covariates including baseline disease characteristics, demographics, lenvatinib exposure, changes in biomarker time profiles, model predicted change from baseline tumor size & change in tumor size time-profiles. Significant (p<0.01) covariates from univariate analysis were added to the model simultaneously & significant predictors retained according to backward exclusion criteria (log likelihood ratio test, p-value = 0.001). Data presented are the predicted change in tumor size estimated using non-linear mixed effects modeling, with Measure Type "Number."
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percent change
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 475
percent change | -0.0523 [-0.0629 to -0.0417]

22. Secondary Outcome: Baseline Tumor Size Estimate for Final Parametric Time to Event PK/PD Model for PFS
Description: Per planned analysis Arms/Groups were combined & PK/PD analysis for PFS was based on lenvatinib & placebo data from this study combined with E7080-G000-303(NCT01321554).Relationship between lenvatinib exposure & PFS was assessed using Kaplan-Meier plots.Parametric survival model(proportional hazard model)with Weibull distribution structure was developed to estimate probability distribution of time from study start to progression as function of covariates including baseline disease characteristics,demographics,lenvatinib exposure,changes in biomarker time profiles,model predicted change from baseline tumor size & change in tumor size time-profiles.Significant(p<0.01)covariates from univariate analysis were added to model simultaneously & significant predictors retained as per backward exclusion criteria(log likelihood ratio test,p-value of 0.001).Data presented are predicted baseline tumor size from the model with Measure Type "Number"estimated using non-linear mixed effects modelling.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: per millimeter (/mm)
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 475
per millimeter (/mm) | -0.00547 [-0.00821 to -0.00273]

23. Secondary Outcome: Input Rate Indirect Effect Model Estimate From Base/Final PK/PD Blood Pressure Model
Description: Per the planned analysis, Arms/Groups were combined and population PK/PD analysis for blood pressure was based on lenvatinib and placebo pooled data from this study combined with study E7080-G000-201 (NCT00784303) & study E7080-G000-303 (NCT01321554). The effect of lenvatinib exposure (AUC) at the time of blood pressure assessment on systolic and diastolic blood pressure was tested as a simultaneous indirect model where lenvatinib AUC was linked to the input rate of the indirect effect model by a linear slope factor function. Based on the results from model development, an indirect PK/PD model with a linear effect of lenvatinib exposure on both systolic and diastolic blood pressure was selected as the base model for subsequent univariate analysis. The data presented are the input rate indirect effect model estimate, with Measure Type "Number." They are population PK/PD model predictions and have been estimated using mixed effects non-linear modeling.
Time Frame: From date of first administration of study drug up to 6 months
Population: For PK/PD analyses of blood pressure, participants received lenvatinib in studies E7080-G000-211, E7080-G000-201 (NCT00784303) and E7080-G000-303 (NCT01321554), with PK information and who had at least one post-baseline evaluation, and participants received placebo in study E7080-G000-303 were included. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: millimeters of mercury per hour
Groups:
- Lenvatinib or Placebo - All Participants: All participants who received lenvatinib 24 mg or 18 mg or placebo, capsule, orally, once daily in a 28-day treatment cycles until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first in studies E7080-G000-303 (NCT01321554), E7080-G000-201 (NCT00784303) and this current study (E7080-G000-211).
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 660
millimeters of mercury per hour | 2.76 [0.978 to 4.54]

24. Secondary Outcome: Drug Effect on Systolic and Diastolic Input Rate Estimates From Base/Final PK/PD Blood Pressure Model
Description: Per the planned analysis, Arms/Groups were combined and population PK/PD analysis for blood pressure was based on lenvatinib and placebo pooled data from this study combined with study E7080-G000-201 (NCT00784303) & study E7080-G000-303 (NCT01321554). The effect of lenvatinib exposure (AUC) at the time of blood pressure assessment on systolic and diastolic blood pressure was tested as a simultaneous indirect model where lenvatinib AUC was linked to the input rate of the indirect effect model by a linear slope factor function. Based on the results from model development, an indirect PK/PD model with a linear effect of lenvatinib exposure on both systolic and diastolic blood pressure was selected as the base model for subsequent univariate analysis. The data presented are the input rate indirect effect model estimate, with Measure Type "Number." They are population PK/PD model predictions and have been estimated using non-linear mixed effects modeling.
Time Frame: From date of first administration of study drug up to 6 months
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: per nanogram*hour per mL*10^6
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 660
per nanogram*hour per mL*10^6
  Drug effect on systolic input rate | 12.0 [10.8 to 13.2]
  Drug effect on diastolic input rate | 21.1 [19.0 to 23.2]

25. Secondary Outcome: Number of Participants With Weight Decrease Stratified by AUC Quartile (Q) Group
Description: Per the planned analysis for this endpoint, Arms/Groups were combined and a population PK/PD analysis of the relationship between lenvatinib exposure and occurrence of the TEAE weight decreased was based on placebo and lenvatinib pooled data from this study combined with study E7080-G000-201 (NCT00784303) and study E7080-G000-303 (NCT01321554). The relationship of occurrence probability of different grades of the TEAE weight decreased and lenvatinib exposure were evaluated by logistic regression model. The logit model was of the form: sum of intercept, of lenvatinib exposure, effects of covariates were explored, and random effects were used to describe between participant variability. Lenvatinib exposure was AUC based on the dose at the time of event. For each TEAE, probabilities of having no TEAE and a CTCAE Version 4.03 Grade 1 (Mild), Grade 2 (Moderate) or Grade 3 (severe or medically significant) TEAE were estimated as a function of lenvatinib or exposure.
Time Frame: Up to 3 years 3 months
Population: For PK/PD analysis of the TEAE weight decreased,participants with DTC who received lenvatinib and placebo from studies E7080-G000-211,E7080-G000-201(NCT00784303)and E7080-G000-303 (NCT01321554)with PK information and who had at least 1 postbaseline safety evaluation were included in analysis.Overall number of participants analyzed signifies participants who were evaluable for outcome measure.Number analyzed signifies participants who were evaluable for this outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Groups:
- Lenvatinib or Placebo - All Participants: All participants received lenvatinib 24 mg or 18 mg or placebo, capsule orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first in studies E7080-G000-303 (NCT01321554), E7080-G000-201 (NCT00784303) and this current study (E7080-G000-211) with available pharmacokinetic data.
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 136
Participants
  AUC Q1; None: number analyzed (Participants) | 135
  AUC Q1; None | 82
  AUC Q1; Grade 1: number analyzed (Participants) | 135
  AUC Q1; Grade 1 | 20
  AUC Q1; Grade 2: number analyzed (Participants) | 135
  AUC Q1; Grade 2 | 29
  AUC Q1; Grade 3: number analyzed (Participants) | 135
  AUC Q1; Grade 3 | 4
  AUC Q2; None: number analyzed (Participants) | 135
  AUC Q2; None | 75
  AUC Q2; Grade 1: number analyzed (Participants) | 135
  AUC Q2; Grade 1 | 17
  AUC Q2; Grade 2: number analyzed (Participants) | 135
  AUC Q2; Grade 2 | 28
  AUC Q2; Grade 3: number analyzed (Participants) | 135
  AUC Q2; Grade 3 | 15
  AUC Q3; None | 74
  AUC Q3; Grade 1 | 18
  AUC Q3; Grade 2 | 33
  AUC Q3; Grade 3 | 11
  AUC Q4; None: number analyzed (Participants) | 135
  AUC Q4; None | 67
  AUC Q4; Grade 1: number analyzed (Participants) | 135
  AUC Q4; Grade 1 | 15
  AUC Q4; Grade 2: number analyzed (Participants) | 135
  AUC Q4; Grade 2 | 37
  AUC Q4; Grade 3: number analyzed (Participants) | 135
  AUC Q4; Grade 3 | 16

26. Secondary Outcome: Number of Participants With Hypertension Stratified by AUC Quartile (Q) Group
Description: Per the planned analysis for this endpoint, Arms/Groups were combined & a population PK/PD analysis of the relationship between lenvatinib exposure & occurrence of the TEAE hypertension was based on placebo & lenvatinib pooled data from this study combined with study E7080-G000-201 (NCT00784303) & study E7080-G000-303 (NCT01321554). The relationship of occurrence probability of different grades of the TEAE hypertension & lenvatinib exposure were evaluated by logistic regression model. The logit model was of the form: sum of intercept, of lenvatinib exposure, effects of covariates were explored, & random effects were used to describe between participant variability. Lenvatinib exposure was AUC based on the dose at the time of event. For each TEAE, probabilities of having no TEAE & a CTCAE Version 4.03 Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (severe or medically significant) or Grade 4 (life-threatening consequences) TEAE were estimated as a function of lenvatinib or exposure.
Time Frame: Up to 3 years 3 months
Population: For PK/PD analysis of the TEAE hypertension,participants with DTC who received lenvatinib and placebo from studies E7080-G000-211,E7080-G000-201(NCT00784303)and E7080-G000-303 (NCT01321554)with PK information and who had at least 1 postbaseline safety evaluation were included in analysis.Overall number of participants analyzed signifies participants who were evaluable for outcome measure.Number analyzed signifies participants who were evaluable for this outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 136
Participants
  AUC Q1; None: number analyzed (Participants) | 135
  AUC Q1; None | 54
  AUC Q1; Grade 1: number analyzed (Participants) | 135
  AUC Q1; Grade 1 | 14
  AUC Q1; Grade 2: number analyzed (Participants) | 135
  AUC Q1; Grade 2 | 37
  AUC Q1; Grade 3: number analyzed (Participants) | 135
  AUC Q1; Grade 3 | 30
  AUC Q1; Grade 4: number analyzed (Participants) | 135
  AUC Q1; Grade 4 | 0
  AUC Q2; None: number analyzed (Participants) | 135
  AUC Q2; None | 48
  AUC Q2; Grade 1: number analyzed (Participants) | 135
  AUC Q2; Grade 1 | 11
  AUC Q2; Grade 2: number analyzed (Participants) | 135
  AUC Q2; Grade 2 | 30
  AUC Q2; Grade 3: number analyzed (Participants) | 135
  AUC Q2; Grade 3 | 47
  AUC Q2; Grade 4: number analyzed (Participants) | 135
  AUC Q2; Grade 4 | 0
  AUC Q3; None | 45
  AUC Q3; Grade 1 | 10
  AUC Q3; Grade 2 | 31
  AUC Q3; Grade 3 | 50
  AUC Q3; Grade 4 | 0
  AUC Q4; None: number analyzed (Participants) | 135
  AUC Q4; None | 51
  AUC Q4; Grade 1: number analyzed (Participants) | 135
  AUC Q4; Grade 1 | 12
  AUC Q4; Grade 2: number analyzed (Participants) | 135
  AUC Q4; Grade 2 | 31
  AUC Q4; Grade 3: number analyzed (Participants) | 135
  AUC Q4; Grade 3 | 40
  AUC Q4; Grade 4: number analyzed (Participants) | 135
  AUC Q4; Grade 4 | 1

27. Secondary Outcome: Number of Participants With Proteinuria Stratified by AUC Quartile (Q) Group
Description: Per the planned analysis for this endpoint, Arms/Groups were combined and a population PK/PD analysis of the relationship between lenvatinib exposure and occurrence of the TEAE proteinuria was based on placebo and lenvatinib pooled data from this study combined with study E7080-G000-201 (NCT00784303) and study E7080-G000-303 (NCT01321554). The relationship of occurrence probability of different grades of the TEAE proteinuria and lenvatinib exposure were evaluated by logistic regression model. The logit model was of the form: sum of intercept, of lenvatinib exposure, effects of covariates were explored, and random effects were used to describe between participant variability. Lenvatinib exposure was AUC based on the dose at the time of event. For each TEAE, probabilities of having no TEAE and a CTCAE Version 4.03 Grade 1 (Mild), Grade 2 (Moderate), or Grade 3 (severe or medically significant) TEAE were estimated as a function of lenvatinib or exposure.
Time Frame: Up to 3 years 3 months
Population: For PK/PD analysis of the TEAE proteinuria,participants with DTC who received lenvatinib and placebo from studies E7080-G000-211,E7080-G000-201(NCT00784303)and E7080-G000-303 (NCT01321554)with PK information and who had at least 1 postbaseline safety evaluation were included in analysis.Overall number of participants analyzed signifies participants who were evaluable for outcome measure.Number analyzed signifies participants who were evaluable for this outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 136
Participants
  AUC Q1; None: number analyzed (Participants) | 135
  AUC Q1; None | 104
  AUC Q1; Grade 1: number analyzed (Participants) | 135
  AUC Q1; Grade 1 | 12
  AUC Q1; Grade 2: number analyzed (Participants) | 135
  AUC Q1; Grade 2 | 13
  AUC Q1; Grade 3: number analyzed (Participants) | 135
  AUC Q1; Grade 3 | 6
  AUC Q2; None: number analyzed (Participants) | 135
  AUC Q2; None | 92
  AUC Q2; Grade 1: number analyzed (Participants) | 135
  AUC Q2; Grade 1 | 7
  AUC Q2; Grade 2: number analyzed (Participants) | 135
  AUC Q2; Grade 2 | 21
  AUC Q2; Grade 3: number analyzed (Participants) | 135
  AUC Q2; Grade 3 | 15
  AUC Q3; None | 72
  AUC Q3; Grade 1 | 16
  AUC Q3; Grade 2 | 32
  AUC Q3; Grade 3 | 16
  AUC Q4; None: number analyzed (Participants) | 135
  AUC Q4; None | 72
  AUC Q4; Grade 1: number analyzed (Participants) | 135
  AUC Q4; Grade 1 | 19
  AUC Q4; Grade 2: number analyzed (Participants) | 135
  AUC Q4; Grade 2 | 34
  AUC Q4; Grade 3: number analyzed (Participants) | 135
  AUC Q4; Grade 3 | 10

28. Secondary Outcome: Number of Participants With Fatigue Stratified by AUC Quartile (Q) Group
Description: Per the planned analysis for this endpoint, Arms/Groups were combined and a population PK/PD analysis of the relationship between lenvatinib exposure and occurrence of the TEAE fatigue was based on placebo and lenvatinib pooled data from this study combined with study E7080-G000-201 (NCT00784303) and study E7080-G000-303 (NCT01321554). The relationship of occurrence probability of different grades of the TEAE fatigue and lenvatinib exposure were evaluated by logistic regression model. The logit model was of the form: sum of intercept, of lenvatinib exposure, effects of covariates were explored, and random effects were used to describe between participant variability. Lenvatinib exposure was AUC based on the dose at the time of event. For each TEAE, probabilities of having no TEAE and a CTCAE Version 4.03 Grade 1 (Mild), Grade 2 (Moderate) or Grade 3 (severe or medically significant) TEAE were estimated as a function of lenvatinib or exposure.
Time Frame: Up to 3 years 3 months
Population: For PK/PD analysis of the TEAE fatigue,participants with DTC who received lenvatinib and placebo from studies E7080-G000-211,E7080-G000-201(NCT00784303)and E7080-G000-303 (NCT01321554)with PK information and who had at least 1 postbaseline safety evaluation were included in analysis.Overall number of participants analyzed signifies participants who were evaluable for outcome measure.Number analyzed signifies participants who were evaluable for this outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 136
Participants
  AUC Q1; None: number analyzed (Participants) | 135
  AUC Q1; None | 75
  AUC Q1; Grade 1: number analyzed (Participants) | 135
  AUC Q1; Grade 1 | 27
  AUC Q1; Grade 2: number analyzed (Participants) | 135
  AUC Q1; Grade 2 | 30
  AUC Q1; Grade 3: number analyzed (Participants) | 135
  AUC Q1; Grade 3 | 3
  AUC Q2; None: number analyzed (Participants) | 135
  AUC Q2; None | 81
  AUC Q2; Grade 1: number analyzed (Participants) | 135
  AUC Q2; Grade 1 | 32
  AUC Q2; Grade 2: number analyzed (Participants) | 135
  AUC Q2; Grade 2 | 17
  AUC Q2; Grade 3: number analyzed (Participants) | 135
  AUC Q2; Grade 3 | 5
  AUC Q3; None | 73
  AUC Q3; Grade 1 | 42
  AUC Q3; Grade 2 | 11
  AUC Q3; Grade 3 | 10
  AUC Q4; None: number analyzed (Participants) | 135
  AUC Q4; None | 79
  AUC Q4; Grade 1: number analyzed (Participants) | 135
  AUC Q4; Grade 1 | 25
  AUC Q4; Grade 2: number analyzed (Participants) | 135
  AUC Q4; Grade 2 | 26
  AUC Q4; Grade 3: number analyzed (Participants) | 135
  AUC Q4; Grade 3 | 5

29. Secondary Outcome: Number of Participants With Diarrhea Stratified by AUC Quartile (Q) Group
Description: Per the planned analysis for this endpoint, Arms/Groups were combined and a population PK/PD analysis of the relationship between lenvatinib exposure and occurrence of the TEAE diarrhea was based on placebo and lenvatinib pooled data from this study combined with study E7080-G000-201 (NCT00784303) and study E7080-G000-303 (NCT01321554). The relationship of occurrence probability of different grades of the TEAE diarrhea and lenvatinib exposure were evaluated by logistic regression model. The logit model was of the form: sum of intercept, of lenvatinib exposure, effects of covariates were explored, and random effects were used to describe between participant variability. Lenvatinib exposure was AUC based on the dose at the time of event. For each TEAE, probabilities of having no TEAE and a CTCAE Version 4.03 Grade 1 (Mild), Grade 2 (Moderate) or Grade 3 (severe or medically significant) TEAE were estimated as a function of lenvatinib or exposure.
Time Frame: Up to 3 years 3 months
Population: For PK/PD analysis of the TEAE diarrhea,participants with DTC who received lenvatinib and placebo from studies E7080-G000-211,E7080-G000-201(NCT00784303)and E7080-G000-303 (NCT01321554)with PK information and who had at least 1 postbaseline safety evaluation were included in analysis.Overall number of participants analyzed signifies participants who were evaluable for outcome measure.Number analyzed signifies participants who were evaluable for this outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 136
Participants
  AUC Q1; None: number analyzed (Participants) | 135
  AUC Q1; None | 55
  AUC Q1; Grade 1: number analyzed (Participants) | 135
  AUC Q1; Grade 1 | 39
  AUC Q1; Grade 2: number analyzed (Participants) | 135
  AUC Q1; Grade 2 | 35
  AUC Q1; Grade 3: number analyzed (Participants) | 135
  AUC Q1; Grade 3 | 6
  AUC Q2; None: number analyzed (Participants) | 135
  AUC Q2; None | 53
  AUC Q2; Grade 1: number analyzed (Participants) | 135
  AUC Q2; Grade 1 | 45
  AUC Q2; Grade 2: number analyzed (Participants) | 135
  AUC Q2; Grade 2 | 29
  AUC Q2; Grade 3: number analyzed (Participants) | 135
  AUC Q2; Grade 3 | 8
  AUC Q3; None | 52
  AUC Q3; Grade 1 | 34
  AUC Q3; Grade 2 | 33
  AUC Q3; Grade 3 | 17
  AUC Q4; None: number analyzed (Participants) | 135
  AUC Q4; None | 56
  AUC Q4; Grade 1: number analyzed (Participants) | 135
  AUC Q4; Grade 1 | 37
  AUC Q4; Grade 2: number analyzed (Participants) | 135
  AUC Q4; Grade 2 | 34
  AUC Q4; Grade 3: number analyzed (Participants) | 135
  AUC Q4; Grade 3 | 8

30. Secondary Outcome: Number of Participants With Nausea Stratified by AUC Quartile (Q) Group
Description: Per the planned analysis for this endpoint, Arms/Groups were combined and a population PK/PD analysis of the relationship between lenvatinib exposure and occurrence of the TEAE nausea was based on placebo and lenvatinib pooled data from this study combined with study E7080-G000-201 (NCT00784303) and study E7080-G000-303 (NCT01321554). The relationship of occurrence probability of different grades of the TEAE nausea and lenvatinib exposure were evaluated by logistic regression model. The logit model was of the form: sum of intercept, of lenvatinib exposure, effects of covariates were explored, and random effects were used to describe between participant variability. Lenvatinib exposure was AUC based on the dose at the time of event. For each TEAE, probabilities of having no TEAE and a CTCAE Version 4.03 Grade 1 (Mild), Grade 2 (Moderate) or Grade 3 (severe or medically significant) TEAE were estimated as a function of lenvatinib or exposure.
Time Frame: Up to 3 years 3 months
Population: For PK/PD analysis of the TEAE nausea,participants with DTC who received lenvatinib and placebo from studies E7080-G000-211,E7080-G000-201(NCT00784303)and E7080-G000-303 (NCT01321554)with PK information and who had at least 1 postbaseline safety evaluation were included in analysis.Overall number of participants analyzed signifies participants who were evaluable for outcome measure.Number analyzed signifies participants who were evaluable for this outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 136
Participants
  AUC Q1; None: number analyzed (Participants) | 135
  AUC Q1; None | 88
  AUC Q1; Grade 1: number analyzed (Participants) | 135
  AUC Q1; Grade 1 | 32
  AUC Q1; Grade 2: number analyzed (Participants) | 135
  AUC Q1; Grade 2 | 14
  AUC Q1; Grade 3: number analyzed (Participants) | 135
  AUC Q1; Grade 3 | 1
  AUC Q2; None: number analyzed (Participants) | 135
  AUC Q2; None | 79
  AUC Q2; Grade 1: number analyzed (Participants) | 135
  AUC Q2; Grade 1 | 36
  AUC Q2; Grade 2: number analyzed (Participants) | 135
  AUC Q2; Grade 2 | 18
  AUC Q2; Grade 3: number analyzed (Participants) | 135
  AUC Q2; Grade 3 | 2
  AUC Q3; None | 83
  AUC Q3; Grade 1 | 37
  AUC Q3; Grade 2 | 14
  AUC Q3; Grade 3 | 2
  AUC Q4; None: number analyzed (Participants) | 135
  AUC Q4; None | 63
  AUC Q4; Grade 1: number analyzed (Participants) | 135
  AUC Q4; Grade 1 | 41
  AUC Q4; Grade 2: number analyzed (Participants) | 135
  AUC Q4; Grade 2 | 29
  AUC Q4; Grade 3: number analyzed (Participants) | 135
  AUC Q4; Grade 3 | 2

31. Secondary Outcome: Number of Participants With Vomiting Stratified by AUC Quartile (Q) Group
Description: Per the planned analysis for this endpoint, Arms/Groups were combined and a population PK/PD analysis of the relationship between lenvatinib exposure and occurrence of the TEAE vomiting was based on placebo and lenvatinib pooled data from this study combined with study E7080-G000-201 (NCT00784303) and study E7080-G000-303 (NCT01321554). The relationship of occurrence probability of different grades of the TEAE vomiting and lenvatinib exposure were evaluated by logistic regression model. The logit model was of the form: sum of intercept, of lenvatinib exposure, effects of covariates were explored, and random effects were used to describe between participant variability. Lenvatinib exposure was AUC based on the dose at the time of event. For each TEAE, probabilities of having no TEAE and a CTCAE Version 4.03 Grade 1 (Mild), Grade 2 (Moderate) or Grade 3 (severe or medically significant) TEAE were estimated as a function of lenvatinib or exposure.
Time Frame: Up to 3 years 3 months
Population: For PK/PD analysis of the TEAE vomiting, participants with DTC who received lenvatinib and placebo from studies E7080-G000-211,E7080-G000-201(NCT00784303)and E7080-G000-303 (NCT01321554)with PK information and who had at least 1 postbaseline safety evaluation were included in analysis. Overall number of participants analyzed signifies participants who were evaluable for outcome measure. Number analyzed signifies participants who were evaluable for this outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib or Placebo - All Participants
Number analyzed (Participants) | 136
Participants
  AUC Q1; None: number analyzed (Participants) | 135
  AUC Q1; None | 106
  AUC Q1; Grade 1: number analyzed (Participants) | 135
  AUC Q1; Grade 1 | 19
  AUC Q1; Grade 2: number analyzed (Participants) | 135
  AUC Q1; Grade 2 | 7
  AUC Q1; Grade 3: number analyzed (Participants) | 135
  AUC Q1; Grade 3 | 3
  AUC Q2; None: number analyzed (Participants) | 135
  AUC Q2; None | 100
  AUC Q2; Grade 1: number analyzed (Participants) | 135
  AUC Q2; Grade 1 | 21
  AUC Q2; Grade 2: number analyzed (Participants) | 135
  AUC Q2; Grade 2 | 11
  AUC Q2; Grade 3: number analyzed (Participants) | 135
  AUC Q2; Grade 3 | 3
  AUC Q3; None | 94
  AUC Q3; Grade 1 | 31
  AUC Q3; Grade 2 | 8
  AUC Q3; Grade 3 | 3
  AUC Q4; None: number analyzed (Participants) | 135
  AUC Q4; None | 86
  AUC Q4; Grade 1: number analyzed (Participants) | 135
  AUC Q4; Grade 1 | 30
  AUC Q4; Grade 2: number analyzed (Participants) | 135
  AUC Q4; Grade 2 | 18
  AUC Q4; Grade 3: number analyzed (Participants) | 135
  AUC Q4; Grade 3 | 1

32. Secondary Outcome: Change From Baseline in the Health-Related Quality of Life (HRQoL) Assessed by European Quality of Life (EuroQol) Five-Dimensional, 3-Level (EQ-5D-3L) Index Score and Visual Analogue Scale (VAS)
Description: The EQ-5D-3L is a health profile questionnaire assessing quality of life along 5 dimensions. Participants rate 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The summed score ranges from 5-15 with "5" corresponding to no problems and "15" corresponding to severe problems in the 5 dimensions. EQ-5D-3L also included an EQ visual analogue scale (VAS) that ranges between 100 (best imaginable health) and 0 (worst imaginable health). Decrease from baseline in EQ-5D-3L signifies improvement. Total index EQ-5D-3L summary score was weighted with a range of -0.594 (worst) to 1.0 (best). EQ-5D-3L also included an EQ health utilities index (HUI) where 1 indicated full health while a score of 0 indicated worst health/death.
Time Frame: Baseline, Week 8, 16, and 24
Population: FAS included all participants randomly assigned to treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lenvatinib 18 mg: Participants initially received lenvatinib 18 mg, capsule, orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first (up to 35 months). To maintain blinded treatment assignment, participants received a total of 4 capsules in the form of one 10-mg capsule and two 4-mg capsules containing lenvatinib and one 10-mg placebo capsule.
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
score on a scale
  EQ-HUI; Baseline | 0.8 (0.17) | 0.8 (0.23)
  EQ-HUI; Change at week 8 | -0.1 (0.19) | 0.0 (0.15)
  EQ-HUI; Change at week 16 | -0.1 (0.20) | -0.1 (0.22)
  EQ-HUI; Change at week 24 | -0.1 (0.17) | -0.1 (0.19)
  EQ-VAS; Baseline | 71.1 (19.12) | 69.2 (21.29)
  EQ-VAS; Change at week 8 | -6.2 (15.71) | -1.4 (19.46)
  EQ-VAS; Change at week 16 | -6.3 (17.08) | -9.8 (17.82)
  EQ-VAS; Change at week 24 | -3.1 (12.95) | -5.1 (23.41)

33. Secondary Outcome: Change From Baseline in the HRQoL Assessed by Functional Assessment of Cancer Therapy-General (FACT-G) Total Score
Description: The FACT-G is a 27-item questionnaire that measures the effect of cancer treatment on quality of life that has four areas of measurements (physical well-being, social/family well-being, emotional well-being and functional well-being). Each item has a 5-point scale response set (0: not at all; 1: a little bit; 2: somewhat; 3: quite a bit; and 4: very much). The FACT-G total score ranges between 0 and 108. Higher score indicates better quality of life.
Time Frame: Baseline, Week 8, 16 and 24
Population: FAS included all participants randomly assigned to treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lenvatinib 24 mg: Participants initially received lenvatinib 24 mg, capsule, orally, once daily in a 28-day treatment cycle until PD, development of unacceptable toxicity, participant requested to discontinue treatment, withdrew consent or lost to follow-up, until the end of the study, or until study termination by the sponsor, whichever occurred first (up to 35 months). To maintain blinded treatment assignment, participants received a total of 4 capsules in the form of two 10-mg capsules and one 4-mg capsule containing lenvatinib and one 4-mg placebo capsule.
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
Number analyzed (Participants) | 75 | 77
score on a scale
  At Baseline | 81.1 (16.18) | 77.8 (16.04)
  Change at Week 8 | -3.0 (12.26) | -1.3 (13.31)
  Change at Week 16 | -4.5 (12.64) | -3.8 (14.75)
  Change at Week 24 | -6.3 (15.49) | -1.5 (16.74)

ADVERSE EVENTS:
Time Frame: From date of first administration of study drug up to 28 days after last dose of study drug up to approximately 3 years 3 months
Arm/Group | Lenvatinib 24 mg | Lenvatinib 18 mg
All-Cause Mortality (participants affected / at risk) | 11/75 | 19/77
Serious Adverse Events (participants affected / at risk) | 26/75 | 35/77
Other Adverse Events (participants affected / at risk) | 75/75 | 76/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib 24 mg (N=75) | Lenvatinib 18 mg (N=77)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Retinal vascular occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (2)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 1 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 2 (3)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (2)
Post-traumatic epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib 24 mg (N=75) | Lenvatinib 18 mg (N=77)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 8 (13)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 3 (8)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (12)
Microcytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 2 (7)
Neutrophilia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (17) | 4 (10)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 2 (4)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (2) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 5 (6) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 5 (5)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid haemorrhage (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (2) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Retinal vascular occlusion (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 18 (27) | 10 (14)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 10 (15) | 13 (21)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Apical granuloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9) | 20 (21)
Dental caries (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 43 (109) | 40 (80)
Dry mouth (Gastrointestinal disorders) | 10 (10) | 9 (11)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 11 (13) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Faeces pale (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 5 (6)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1) | 2 (5)
Glossodynia (Gastrointestinal disorders) | 2 (4) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lip oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 31 (52) | 28 (36)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 3 (5)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 5 (5) | 3 (4)
Oral pain (Gastrointestinal disorders) | 6 (12) | 6 (8)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 16 (25) | 22 (50)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 6 (6) | 4 (4)
Vomiting (Gastrointestinal disorders) | 15 (22) | 13 (21)
Asthenia (General disorders) | 18 (34) | 21 (51)
Axillary pain (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (5) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Early satiety (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 2 (2)
Facial pain (General disorders) | 1 (1) | 2 (3)
Fatigue (General disorders) | 30 (60) | 28 (56)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 2 (3) | 1 (3)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (2) | 1 (2)
Induration (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 4 (5) | 3 (3)
Malaise (General disorders) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3) | 8 (11)
Oedema (General disorders) | 0 (0) | 2 (3)
Oedema peripheral (General disorders) | 16 (25) | 12 (19)
Pain (General disorders) | 3 (3) | 4 (6)
Pyrexia (General disorders) | 4 (4) | 7 (9)
Temperature intolerance (General disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (4)
Cystitis (Infections and infestations) | 2 (3) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (2) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 4 (5)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (5) | 2 (3)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (4)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (3)
Pneumonia (Infections and infestations) | 3 (3) | 3 (4)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (4) | 5 (6)
Tooth abscess (Infections and infestations) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 1 (2)
Tracheitis (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (8)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (20) | 9 (14)
Amylase increased (Investigations) | 4 (21) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 14 (21) | 9 (17)
Bacterial test positive (Investigations) | 1 (1) | 0 (0)
Biopsy prostate normal (Investigations) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3)
Blood bilirubin increased (Investigations) | 4 (5) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 1 (2)
Blood cholesterol increased (Investigations) | 5 (6) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 3 (7)
Blood creatinine increased (Investigations) | 4 (5) | 6 (8)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (3) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 2 (2)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (2)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 8 (22) | 5 (7)
Electrocardiogram ST-T segment abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (3) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (8)
Glucose urine present (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 7 (21) | 6 (11)
Lymphocyte count decreased (Investigations) | 3 (5) | 7 (9)
Platelet count decreased (Investigations) | 5 (8) | 5 (16)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Tracheal aspiration procedure (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 2 (2)
Troponin I increased (Investigations) | 1 (1) | 1 (1)
Urine ketone body present (Investigations) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 30 (62) | 34 (67)
Weight increased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 2 (2) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 26 (38) | 22 (40)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (7) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8) | 5 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (10)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (10) | 12 (31)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (16) | 6 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (7) | 10 (14)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (8) | 6 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (45) | 22 (39)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (17) | 12 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (7)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 15 (25)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (25) | 17 (33)
Neck pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 11 (15)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (19) | 11 (17)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (7)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 2 (2)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 11 (14) | 6 (8)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (6) | 5 (7)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 19 (24) | 17 (29)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (4) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 4 (5)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 4 (5) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 4 (4) | 3 (4)
Vocal cord paralysis (Nervous system disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 7 (7) | 4 (4)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (7) | 6 (8)
Irritability (Psychiatric disorders) | 1 (2) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Thermophobia (Psychiatric disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (4)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Haematuria (Renal and urinary disorders) | 3 (5) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 35 (169) | 26 (93)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 19 (24)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 20 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 13 (16)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (15)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (9)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (6)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 26 (48) | 22 (45)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 6 (10) | 4 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 44 (127) | 40 (91)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 6 (7)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Toxic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT02702388/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT02702388/SAP_001.pdf